CLINICAL TRIAL: NCT02142673
Title: The Impact of Different Filling Pressures in Operative Outpatient Hysteroscopy on the Procedure Success Rates and Associated Pain. A Randomized Double Blind Controlled Trial
Brief Title: The Impact of Different Filling Pressures in Operative Outpatient Hysteroscopy on the Procedure Success Rates and Associated Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Hyst 2
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Hysteroscopy
Keywords: Operative hysteroscopy; Filling pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Filling pressure 80 (Active Comparator): The hysteroscope filling pressure will be 80mm Hg
  Interventions: Device: Filling pressure 80
- Filling pressure 60 (Active Comparator): The hysteroscope filling pressure will be to 50mm Hg
  Interventions: Device: Filling pressure 60
- Filling pressure 40 (Active Comparator): The hysteroscope filling pressure will be to 40mm Hg
  Interventions: Device: Filling pressure 40

INTERVENTIONS:
Device: Filling pressure 80 — The hysteroscope filling pressure will be 80mm Hg
  Arms: Filling pressure 80
Device: Filling pressure 60 — The hysteroscope filling pressure will be reduced to 50mm Hg
  Arms: Filling pressure 60
Device: Filling pressure 40 — The hysteroscope filling pressure will be 40mm Hg
  Arms: Filling pressure 40

SUMMARY:
The study aims to compare different filling pressures in operative outpatient hysteroscopy. Women will be divided into 3 groups. The hysteroscope will be introduced in the uterine cavity. Saline will be used as the distension medium and the pressure will be 80mm Hg in group1, 60mm Hg in group 2 and 40mmHg in group 3.

DETAILED DESCRIPTION:
240 women will be randomly divided into 3 groups, each containing 80 women. Randomisation will be performed using a computer generated random numbers and sealed envelopes.

Full history will be taken followed by general and local examination. One hour before the procedure all women will receive diclofenac 100mg (Voltaren@ Novartis Switzerland). The procedure will be done in the lithotomy position. Hysteroscopy will be done using a 5mm outer diameter continuous flow hysteroscope with a French working channel and a 30 degrees direction of view provided by Techno GmbH and CO. The hysteroscope will be introduced using the vaginoscopy technique, in which no speculum will be used. The cervix will be detected and the external os will be identified using the hysteroscope. The hysteroscope will be introduced in the uterine cavity. Saline will be used as the distension medium and the pressure will be 80mm Hg in group1, 60mm Hg in group 2 and 40 mmHg in group 3. Randomisation will be double blind, neither the operator nor the patient will know the pressure during the procedure, a third party will set the pressure according to the computer generated random numbers. If the procedure cannot be completed, the operator will ask for the pressure to be adjusted to 80mm Hg, which is the usual pressure used in Cairo university hospitals, or more if needed. In this case the operator will document in the data collection form that the procedure could not be completed with the pre-set pressure.

The anterior wall, posterior wall and tubal ostea will be visualised, any polyps, adhesions septa, congenital malformations or submucous fibroids will be noted. Endometrial biopsy will be taken using a semi-rigid, double action oval serrated biopsy forceps 40cm 50Charr Tecchno medical GmbH. The used scissor will be a single action semi-rigid rounded tip scissors Tecchno medical GmbH.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Indication to have an operative outpatient hysteroscopy like endometrial polyp, need for endometrial biopsy, intrauterine adhesions, intra uterine device (IUD) retrieval or intrauterine septum resection.
* Consents to participate in the study

Exclusion Criteria:

* Premenstrual and mid-menstrual patients.
* Patients with missed periods.
* Patients with known cardiac disease.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2014-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Completing the procedure with the allocated pressure | 30 minutes after starting the procedure
  The operator will document if he is able to complete the operative procedure with the allocated pressure. If the operator is not able to operate with the allocation pressure, he will document that the procedure cannot be completed with the current pressure and will ask for the filling pressure to be adjusted

SECONDARY OUTCOMES:
Pain perception during the procedure | 10 minutes after starting the procedure
  Pain will be assessed using a visual analogue scale 10 minutes after starting the procedure
Pain perception after the procedure | 30 minutes after completing the procedure
  Pain will be assessed using a visual analogue scale 30 minutes after completing the procedure

CONTACTS AND LOCATIONS:
Overall Officials: AbdelGany MA Hassan, MRCOG, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

REFERENCES:
- [Background] Sharma JB, Aruna J, Kumar P, Roy KK, Malhotra N, Kumar S. Comparison of efficacy of oral drotaverine plus mefenamic acid with paracervical block and with intravenous sedation for pain relief during hysteroscopy and endometrial biopsy. Indian J Med Sci. 2009 Jun;63(6):244-52. PMID 19602758
- [Background] van Dongen H, de Kroon CD, Jacobi CE, Trimbos JB, Jansen FW. Diagnostic hysteroscopy in abnormal uterine bleeding: a systematic review and meta-analysis. BJOG. 2007 Jun;114(6):664-75. doi: 10.1111/j.1471-0528.2007.01326.x. PMID 17516956
- [Background] O'Flynn H, Murphy LL, Ahmad G, Watson AJ. Pain relief in outpatient hysteroscopy: a survey of current UK clinical practice. Eur J Obstet Gynecol Reprod Biol. 2011 Jan;154(1):9-15. doi: 10.1016/j.ejogrb.2010.08.015. PMID 20926175
- [Background] Shahid A, Pathak M, Gulumser C, Parker S, Palmer E, Saridogan E. Optimum uterine filling pressure for outpatient diagnostic hysteroscopy: a double-blind, randomized controlled trial. Reprod Biomed Online. 2014 Jan;28(1):86-91. doi: 10.1016/j.rbmo.2013.07.018. Epub 2013 Sep 14. PMID 24262433
- [Derived] Haggag H, Hassan A, Wahba A, Joukhadar R. A randomized double-blind controlled trial of different filling pressures in operative outpatient hysteroscopy. Int J Gynaecol Obstet. 2017 Oct;139(1):55-60. doi: 10.1002/ijgo.12247. Epub 2017 Jul 25. PMID 28653328